CLINICAL TRIAL: NCT06462287
Title: PILOT STUDY OF THE EFFECT OF A SUBSTANCE P ANTAGONIST, APREPITANT, ON THE SECRETION OF ALDOSTERONE IN PATIENTS WITH OBSTRUCTIVE SLEEP APNEA SYNDROME AND ARTERIAL HYPERTENSION
Brief Title: EFFECT OF A SUBSTANCE P ANTAGONIST ON THE SECRETION OF ALDOSTERONE IN PATIENTS WITH OBSTRUCTIVE SLEEP APNEA SYNDROME AND ARTERIAL HYPERTENSION
Acronym: APHOS3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/0431/HP
Record Dates: First submitted 2024-06-04; First posted 2024-06-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aprepitant (Experimental)
  Interventions: Drug: Aprepitant 125 and 80Mg Oral Capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant 125 and 80Mg Oral Capsule — Aprepitant 1 oral capsule time a day for 4 days (First day: 125 mg and the 3 last days: 80 mg)
  Arms: Aprepitant
Drug: Placebo — Placebo:1 oral capsule time a day for 4 days
  Arms: Placebo

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is associated with hyperaldosteronism with elevated plasma aldosterone/renin ratio, the physiopathological mechanism of which remains uncertain. This hyperaldosteronism contributes to the development of arterial hypertension and cardiovascular complications observed in patients with OSA, in particular by increasing arterial stiffness and heart rate variability. The frequent association of OSA with obesity with metabolic syndrome suggests that excess weight could be responsible for stimulation of aldosterone secretion independent of the renin/angiotensin system. Several studies indicate in particular that the production of mineralocorticoids by the adrenals could be activated by various adipocyte secretion products such as leptin and certain fatty acids after oxidation in the liver. In addition, a recent study showed that basal aldosterone secretion is also controlled by substance P released within the adrenal tissue itself by nerve fibers belonging to the splanchnic contingent. Thus, the oral administration of aprepitant, an antagonist of the substance P receptor (NK1 receptor), to healthy volunteers induces a reduction of approximately 30% in the overall secretion of aldosterone assessed by measuring aldosteronemia and 24-hour aldosteronuria. To the extent that OSA causes sympathetic hypertonia, the hypothesis is that the associated hyperaldosteronism could result from activation of the nervous control of aldosterone secretion, involving substance P and the NK1 receptor. If this is indeed the case, the administration of aprepitant to patients with OSA should result in a significant reduction in aldosteronemia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with severe obstructive sleep apnea syndrome (OSAS) defined by an apnea and hypopnea index (AHI) ≥ 30/h on polysomnography or ventilatory polygraphy (requiring continuous positive airway pressure).
2. Subject with essential hypertension treated medically or by lifestyle and dietary measures or newly diagnosed (defined by SBP ≥ 140 and/or DBP ≥ 90 mmHg according to current SFHTA-HAS recommendations).
3. Patient's agreement to replace diuretics with another neutral antihypertensive treatment (which does not interfere with the renin-angiotensin system), to stop consuming licorice and its derivatives, 7 to 10 days before taking the treatment. experimental and throughout the study (if applicable)

Exclusion Criteria:

1. Minor subject or subject aged over 75 years
2. Criteria relating to associated pathologies leading to particular risks:

   * Subject presenting excessive daytime sleepiness with contraindication to driving (Epworth score > 16)
   * Uncontrolled severe cardiovascular disease: myocardial infarction or stroke in the last 6 months, unstable angina, significant valvular heart disease, heart failure (≥ class II of the NYHA classification), uncontrolled cardiac arrhythmia or significant conduction abnormalities. Knowledge of chronic renal insufficiency defined by a glomerular filtration rate < 60 mL/min/1.73m2 for more than 3 months) or moderate hepatic insufficiency defined by ALT and/or AST transaminases > 3N)
   * Epilepsy
   * Known acute infections linked to HIV, HBV or HCV
   * Active cancer currently being treated
3. Contraindications to placebo and aprepitant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-04-19 (Estimated); Study Completion 2026-04-19 (Estimated)

PRIMARY OUTCOMES:
Rate of aldosterone secretion | Immediately after the intervention/procedure/surgery
  Measurement of 24-hour aldosteronuria before and after the administration of an NK1 receptor antagonist (aprepitant) or placebo in patients suffering from obstructive sleep apnea syndrome (OSAS) and arterial hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rouen, Rouen, France, France

IPD SHARING:
Plan to Share IPD: No